CLINICAL TRIAL: NCT03394508
Title: The Safety and Efficacy of Intralymphatic Immunotherapy in Pollen Allergic Adolescents and Young Adults With Asthma: A Randomized Placebo-controlled Trial
Brief Title: The Safety and Efficacy of Intralymphatic Immunotherapy in Pollen Allergic Adolescents and Young Adults With Asthma
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Gunilla Hedlin, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DNR 2012/701 EPN Lund
Record Dates: First submitted 2017-12-06; First posted 2018-01-09 (Actual); Results first posted 2020-09-28 (Actual); Last update posted 2020-09-28 (Actual); Status verified 2020-09

CONDITIONS: Rhinitis; Asthma; Allergy
MeSH Terms: conditions — Rhinitis; Asthma; Hypersensitivity | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): ALK diluent 0,3% human albumin'
  Interventions: Drug: ALK diluent 0,3% human albumin
- Active treatment (Experimental): Intervention: Drug ALK Alutard birch or 5-grasses. Grass pollen suspension or birch pollen suspension
  Interventions: Drug: ALK Alutard birch or 5-grasses

INTERVENTIONS:
Drug: ALK Alutard birch or 5-grasses — Intralymphatic injection with 1000 units. 3 injections with 4-5 weeks interval (0,1 ml) and one additional booster injection with 1000 units before the second pollen season.
  Other Names: ALK Alutard birch pollen or ALK Alutard grass pollen
  Arms: Active treatment
Drug: ALK diluent 0,3% human albumin — Intralymphatic injection with 0.1 ml. 3 injections with 4-5 weeks interval
  Other Names: Human albumin
  Arms: Placebo

SUMMARY:
The study evaluates the safety and efficacy of intralymphatic allergen-specific immunotherapy given to adolescents and young adults who are allergic to grass or birch pollen and have mild or moderate asthma. Patients will be treated with three intralymphatic injections; 1000 SQ-U x3 with 4-5 weeks interval, or placebo with 4-5 weeks interval. The patients receiving treatment will be given a fourth injection one year after the initial injections. The study is conducted in collaboration between Professor Lars Olof Cardell (ENT), prof Gunilla Hedlin (Pediatrics) and prof Marianne van Hage (Immunology)".

DETAILED DESCRIPTION:
30 patients with seasonal allergic rhinitis due to birch or grass pollen are included. Study subjects are randomized to intralymphatic injections with placebo or ALK Alutard 5-grasses / birch or placebo. The patients receiving treatment will be given a fourth injection one year after the initial injections.

ELIGIBILITY:
Inclusion Criteria:

* Allergic rhinitis due to grass or birch pollen
* Mild to moderate asthma with a positive methacholine challenge
* Accepted and signed informed consent.

Exclusion Criteria:

* Previously subcutaneous immunotherapy (SCIT) with total symptom relief.
* Previously SCIT but no symptom improvement at all.
* Sensitizations to house dust mite or furry animals, with ongoing exposure and symptoms.
* Severe atopic dermatitis.
* Patients with significant diseases other than allergic rhinitis. A significant disease is defined as a disease which in the opinion of the investigator may either put the patient at risk because of participation in the study or a disease which may influence the results of the study or the patient's ability to participate in the study.
* Patients with a respiratory tract infection in the past 4 weeks prior to Visit 2.
* Pregnant or nursing women or women of childbearing potential not using a medically approved means of contraception (i.e., oral contraceptives, intrauterine devices, diaphragm, or subdermal implants).
* Known autoimmune or collagen disease
* Cardiovascular disease
* Hepatic disease
* Known renal insufficiency
* Cancer
* Hematologic disease
* Chronic infectious disease
* Any medication with a possible side-effect of interfering with the immune response
* Previous immuno- or chemotherapy
* Disease or conditions rendering the treatment of anaphylactic reactions difficult (symptomatic coronary heart diseases, severe arterial hypertension and treatment with β-blockers)
* Major metabolic disease
* Known or suspected allergy to the study product
* Obesity with BMI > 30 since subcutaneous fat makes ultrasound imaging of lymph nodes harder which may risk the correct placement of injection.
* Patients who, in the opinion of the investigator, abuse alcohol or drugs within 2 years prior to Visit 1.
* Patients who have taken an investigational drug within 1 month or six half lives, whichever is greater, prior to Visit 1.
* Mental incapability of coping with the study
* Withdrawal of informed consent

Ages: 16 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Patterson AM, Bonny AE, Shiels WE 2nd, Erwin EA. Three-injection intralymphatic immunotherapy in adolescents and young adults with grass pollen rhinoconjunctivitis. Ann Allergy Asthma Immunol. 2016 Feb;116(2):168-70. doi: 10.1016/j.anai.2015.11.010. Epub 2015 Dec 17. No abstract available. PMID 26706294
- [Background] Witten M, Malling HJ, Blom L, Poulsen BC, Poulsen LK. Is intralymphatic immunotherapy ready for clinical use in patients with grass pollen allergy? J Allergy Clin Immunol. 2013 Nov;132(5):1248-1252.e5. doi: 10.1016/j.jaci.2013.07.033. Epub 2013 Sep 13. No abstract available. PMID 24035151
- [Background] Hylander T, Latif L, Petersson-Westin U, Cardell LO. Intralymphatic allergen-specific immunotherapy: an effective and safe alternative treatment route for pollen-induced allergic rhinitis. J Allergy Clin Immunol. 2013 Feb;131(2):412-20. doi: 10.1016/j.jaci.2012.10.056. PMID 23374268
- [Background] Senti G, Crameri R, Kuster D, Johansen P, Martinez-Gomez JM, Graf N, Steiner M, Hothorn LA, Gronlund H, Tivig C, Zaleska A, Soyer O, van Hage M, Akdis CA, Akdis M, Rose H, Kundig TM. Intralymphatic immunotherapy for cat allergy induces tolerance after only 3 injections. J Allergy Clin Immunol. 2012 May;129(5):1290-6. doi: 10.1016/j.jaci.2012.02.026. Epub 2012 Mar 30. PMID 22464647
- [Result] Hylander T, Larsson O, Petersson-Westin U, Eriksson M, Kumlien Georen S, Winqvist O, Cardell LO. Intralymphatic immunotherapy of pollen-induced rhinoconjunctivitis: a double-blind placebo-controlled trial. Respir Res. 2016 Jan 27;17:10. doi: 10.1186/s12931-016-0324-9. PMID 26817454

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four patients were removed or left the study before analysis of results; 3 patients (active group) were excluded after the first treatment period because of deviations from the treatment protocol, and 1 patient (placebo) left the study after the first treatment period, before the follow-up
Groups:
- Active Treatment: Intervention: Drug ALK Alutard birch or 5-grasses. Grass pollen suspension or birch pollen suspension
  ALK Alutard birch or 5-grasses: Intralymphatic injection with 1000 units. 3 injections with 4-5 weeks interval and a booster injection with 1000 units before the second pollen season
Period: Overall Study
Arm/Group | Placebo | Active Treatment
Started | 13 | 17
Completed | 12 | 14
Not Completed | 1 | 3
Not completed — Protocol Violation | 0 | 3
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Active Treatment: Intervention: Drug ALK Alutard birch or 5-grasses Grass pollen suspension or birch pollen suspension.
  ALK Alutard birch or 5-grasses: Intralymphatic injection with 1000 units. 3 injections with 4-5 weeks interval and a booster injection with 1000 units before the second pollen season.
- Total: Total of all reporting groups
Arm/Group | Placebo | Active Treatment | Total
Number analyzed (Participants) | 13 | 17 | 30
Age, Continuous [Median (Full Range); unit: years] — Population: Four patients were removed or left the study before analysis of results; 3 patients (active group) were excluded after the first treatment period because of deviations from the treatment protocol, and 1 patient (placebo) left the study after the first treatment period, before the follow-up
  years
    number analyzed (Participants) | 12 | 14 | 26
    (all) | 18 [16 to 36] | 19.5 [16 to 42] | 19 [16 to 42]
Age, Customized [Median (Full Range); unit: years] — Population: Four patients were removed or left the study before analysis of results; 3 patients (active group) were excluded after the first treatment period because of deviations from the treatment protocol, and 1 patient (placebo) left the study after the first treatment period, before the follow-up.
  years
    Age: number analyzed (Participants) | 12 | 14 | 26
    Age | 18 [16 to 36] | 19.5 [16 to 42] | 19 [16 to 42]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Four patients were removed or left the study before analysis of results; 3 patients (active group) were excluded after the first treatment period because of deviations from the treatment protocol, and 1 patient (placebo) left the study after the first treatment period, before the follow-up.
  Participants
    number analyzed (Participants) | 12 | 14 | 26
    Female | 2 | 8 | 10
    Male | 10 | 6 | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Sweden | 13 | 17 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change in Symptoms Score After Nasal Allergen Challenge
Description: 0,1 ml of ALK Aquagen birch or timothy 10 000 SQU/ml is deposited in each nostril and allergy symptoms are recorded. Symptoms during NPTs were scored according to the Lebel scoring scale. Symtom scores at 5, 15, and 30 minutes after nasal administration of the allergenextract were summed to represent the symptom-score at each nasal challenge (at inclusion, 12 months after inclusion and for the active patients 24 months after inclusion). The scoring system identifies nasal, eye, and ear symptoms: rhinorrhea, nasal pruritus, nasal congestion, ocular pruritus, watery eyes, and itchy ears, each graded on a scale from 0 to 3 points, and a total score was summarized after subtracting the starting score (min score is 0 and maximum score is 54 + the number of sneezes). Higher scores mean worse outcome.
Time Frame: At inclusion (pre-treatment), 12 months after inclusion (after first pollen season) and for the active treated patients 24 months after inclusion (after the second pollen season).
Population: Patients were injected 3 times before the start of the first pollen season. The study was unblinded at a follow-up visit after the end of the first season. Active patients returned for a booster injection (1000 SQ-U) before the second season and performed a new follow-up. Eleven patients (6 active, 5 placebo) did not have full analysis data sets.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Active Treatment: Intervention: Drug ALK Alutard birch or 5-grasses Grass pollen suspension or birch pollen suspension
  ALK Alutard birch or 5-grasses: Intralymphatic injection with 1000 units. 3 injections with 4-5 weeks interval and an additional booster injection with 1000 units before the second pollen season.
Arm/Group | Placebo | Active Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  After the first pollen season: number analyzed (Participants) | 11 | 13
  After the first pollen season | -5 [-9 to 5] | -4 [-12 to 4]
  After the second season compared to pre-treatment: number analyzed (Participants) | 0 | 11
  After the second season compared to pre-treatment |  | -1 [-7 to 2]

2. Secondary Outcome: Change on Visual Analogue Scale (VAS
Description: Treatment effect was evaluated by asking the patients to compare their allergic symptoms during the last pollen season with the pollen season before treatment on a visual analogue scale ranging from 0 (unchanged symptoms, no improvement) to 10 (total symptom relief, complete recovery).
Time Frame: as for outcome 1
Population: 4 left the study before analysis of results; 3 active were excluded after the first treatment period because of deviations from the treatment protocol, and 1 placebo left the study after the first treatment period, before the follow-up. 11 patients (6 active, 5 placebo) did not have full analysis data sets, see limitations section for details.
Measure: Median (Full Range); unit: score on a scale
Groups:
- Placebo: ALK diluent 0,3% human albumin'
  ALK diluent 0,1 ml human albumin: Intralymphatic injection. 3 injections with 4-5 weeks interval.
- Active Treatment: Intervention: Drug ALK Alutard birch or 5-grasses Grass pollen suspension or birch pollen suspension.
  ALK Alutard birch or 5-grasses: Intralymphatic injection with 1000 units. 3 injections with 4-5 weeks interval and an additional booster injection with 1000 units before the second pollen season.
Arm/Group | Placebo | Active Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  After first season | 3.5 [0 to 8.5] | 5.5 [0 to 9.1]
  After second season compared to pre-treatment: number analyzed (Participants) | 0 | 12
  After second season compared to pre-treatment |  | 6.9 [0 to 9.5]

3. Secondary Outcome: Change in Quality of Life
Description: Difference before and after treatment in Quality of Life. Quality of life was assessed using the Juniper Asthma Quality of Life Questionnaire, giving a score ranging from 1 to 7, and a change in score of 0.5 points is considered clinically relevant. Lower value is considered worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Placebo | Active Treatment
Number analyzed (Participants) | 12 | 14
units on a scale
  After first season: number analyzed (Participants) | 12 | 12
  After first season | 0.17 [-2 to 2.1] | 0.3 [-0.5 to 1.1]
  After second season compared to pre-treatment: number analyzed (Participants) | 0 | 11
  After second season compared to pre-treatment |  | 0.13 [-1.3 to 1]

4. Secondary Outcome: Change in Allergen-specific Serum Immunoglobulin E (IgE) Levels Compared to Before Treatment
Description: Allergen-specific IgE levels were measured by ImmunoCAP (Thermo Scientific, Uppsala, Sweden) for birch (t3) and timothy grass (g6) pollen according to the manufacturer's instructions. A cutoff level ≥ 0.35 kUA/L was considered positive.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: units on a scale IgE:Kua/L
Groups:
- Placebo: ALK diluent 0,3% human albumin'
  ALK diluent 0.1 ml human albumin: Intralymphatic injection. 3 injections with 4-5 weeks interval
Arm/Group | Placebo | Active Treatment
Number analyzed (Participants) | 12 | 14
units on a scale IgE:Kua/L
  IgE after first season | -0.5 [-370 to 70] | 10.5 [-50 to 116]
  IgE after second season compared to pre-treatment: number analyzed (Participants) | 0 | 13
  IgE after second season compared to pre-treatment |  | 0 [-111 to 83]

5. Secondary Outcome: Change in Asthma Symptom Scores
Description: Asthma control 4 weeks before follow-up was estimated with the asthma control test. The score is based on a questionnaire with 5 questions concerning the patients asthma. Each question can be given a score from 1 to 5 points. The answers for each question is added together, where a minimum score of 5 and a maximum score of 25 can be obtained. Higher scores indicate improved outcome and a score of 19 or less suggests poorly controlled asthma.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Placebo | Active Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  After the first pollen seasonllen season | 0 [-7 to 4] | 0 [-5 to 3]
  After second season compared to pre-treatment: number analyzed (Participants) | 0 | 14
  After second season compared to pre-treatment |  | 1.5 [-10 to 4]

6. Secondary Outcome: Change in Pulmonary Function Measurement (Spirometry)
Description: FEV1 were measured according to international guidelines and results presented in % of predicted values according to the patients height, gender, age and weight.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: percent predicted FEV1
Arm/Group | Placebo | Active Treatment
Number analyzed (Participants) | 12 | 14
percent predicted FEV1
  After first season: number analyzed (Participants) | 11 | 14
  After first season | -3 [-27 to 4] | 1 [-15 to 14]
  After second season compared to pre-treatment: number analyzed (Participants) | 0 | 12
  After second season compared to pre-treatment |  | -5.5 [-32 to 8]

7. Secondary Outcome: Changes in Airway Inflammation Assessed by Exhaled Nitric Oxide
Description: Nitric oxide in exhaled air, p.p.b. were measured according to international guidelines, and higher values indicate worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: parts per billion (ppb)
Arm/Group | Placebo | Active Treatment
Number analyzed (Participants) | 12 | 14
parts per billion (ppb)
  After first season: number analyzed (Participants) | 11 | 14
  After first season | -5 [-52 to 19] | 1 [-27 to 13]
  After second season compared to pre-treatment: number analyzed (Participants) | 0 | 12
  After second season compared to pre-treatment |  | -2.5 [-28 to 28]

8. Secondary Outcome: Change in Symptom and Medication-score
Description: Modified Symptom scores and Medication score were calculated taking into account the frequency: daily (4 points); every second day (3 points); 1 to 3 days per week (2 points); occasionally (1 point); never (0 points), for the following symptoms: blocked nose, rhinorrhea, fatigue, sneezing, and asthma symptoms, and for the following medications used: local and systemic antihistamines, nasal steroids, asthma medication, and eye drops. A minimum score of 0 and a maximum score of 20 points for symptoms and 16 points for medication could be obtained. Higher values indicate worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Placebo | Active Treatment
Number analyzed (Participants) | 12 | 14
score on a scale
  Symptom score after first season: number analyzed (Participants) | 9 | 11
  Symptom score after first season | -3 [-7 to 0] | -4 [-13 to 2]
  Medication score after first season: number analyzed (Participants) | 9 | 11
  Medication score after first season | -2 [-4 to 3] | -2 [-11 to 2]
  Symptom score after second season: number analyzed (Participants) | 0 | 10
  Symptom score after second season |  | -5 [-15 to 0]
  Medication score after second season: number analyzed (Participants) | 0 | 10
  Medication score after second season |  | -3 [-12 to -1]

9. Secondary Outcome: Changes in Response to a Bronchial Challenge With Methacholine
Description: Methacholine challenge to test the bronchial hyperresponsiveness in the airways of the included subjects. The subject will inhale increasing doses of methacholine. Spirometry is performed before and between each inhalation. The cumulative dose of methacholine needed to elicit at 20% decrease in FEV1 (PD20) is reported. Lower values indicate worse outcome.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: units on a scale PD20
Arm/Group | Placebo | Active Treatment
Number analyzed (Participants) | 12 | 14
units on a scale PD20
  After the first pollen season: number analyzed (Participants) | 11 | 14
  After the first pollen season | -5 [-150 to 203] | 23 [-131 to 278]
  After the second pollen season compared to pre-tre: number analyzed (Participants) | 0 | 11
  After the second pollen season compared to pre-tre |  | 53 [-34 to 489]

10. Secondary Outcome: Change in Allergen-specific Serum Immunoglobulin (Ig) G and Ig4 Levels Compared to Before Treatment
Description: Allergen-specific IgG and IgG4 level was measured by ImmunoCAP (Thermo Scientific, Uppsala, Sweden) for birch (t3) and timothy grass (g6) pollen according to the manufacturer's instructions. A cutoff 2 mg/L for IgG and 0.05 mg/L for IgG4 was considered positive.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: mg/L
Arm/Group | Placebo | Active Treatment
Number analyzed (Participants) | 12 | 14
mg/L
  IgG after first season | -0.25 [-1 to 1] | 0.6 [-1.3 to 2.9]
  IgG4 after first season | 0.03 [-0.76 to 0.08] | 0.12 [-0.73 to 2]
  IgG after second season compared to pre-treatment: number analyzed (Participants) | 0 | 13
  IgG after second season compared to pre-treatment |  | -0.2 [-2.5 to 4]
  IgG4 after second season compared to pre-treatment: number analyzed (Participants) | 0 | 13
  IgG4 after second season compared to pre-treatment |  | 0 [-0.3 to 0.69]

ADVERSE EVENTS:
Time Frame: Within 24 hours after each injection, up to 24 months for patients receiving active treatment and up to 12 months for patients receiving placebo.
Groups:
- Placebo: ALK diluent 0,3% human albumin'
  ALK diluent 0.1 ml human albumin: Intralymphatic injection with 1000 units. 3 injections with 4-5 weeks interval
- Active Treatment: Intervention: Drug ALK Alutard birch or 5-grasses Grass pollen suspension or birch pollen suspension
  ALK Alutard birch or 5-grasses: Intralymphatic injection with 1000 units. 3 injections with 4-5 weeks interval and an additional booster injection before the second pollen season.
Arm/Group | Placebo | Active Treatment
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/13 | 2/17
Other Adverse Events (participants affected / at risk) | 5/13 | 13/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Active Treatment (N=17)
Generalized urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — One patient was diagnosed with Sarcoidosis 3 months after the booster injection.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=13) | Active Treatment (N=17)
Pain (Nervous system disorders) | 1 | 4
Redness (Skin and subcutaneous tissue disorders) | 1 | 8
Itchyness (Skin and subcutaneous tissue disorders) | 0 | 9
Swollen locally around injection site (Skin and subcutaneous tissue disorders) | 1 | 8
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tiredness (Nervous system disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 — The patient reported worsened eczema after the first treatment period and declined the booster dose

LIMITATIONS AND CAVEATS:
a=active,p=placebo:No booster dose and no follow-up (1a), No NPTs before (1a) and at follow up (1a, 1p), No methacholine, quality of life in the second follow-up (1a). No symptoms and medication scores (3a, 3p), No spirometry at follow-up (1a,1p).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT03394508/Prot_SAP_000.pdf